CLINICAL TRIAL: NCT05018507
Title: NavOne - Variations in Osteoarthritic Knee Laxity Between Individuals and Populations
Brief Title: Variations in Osteoarthritic Knee Laxity Between Individuals and Populations
Acronym: NavOne
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021ORT117
Record Dates: First submitted 2021-06-16; First posted 2021-08-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- total knee arthroplasty patients: data collection only
  Interventions: Other: Data collection only

INTERVENTIONS:
Other: Data collection only — No intervention, just data collection from system machines

SUMMARY:
Severe osteoarthritis of the knee is a condition associated with severe pain, disability and a loss of independence. The most definitive method of surgical treatment for this condition is total knee arthroplasty (TKA). Total knee arthroplasty aims to provide new metallic bearing surfaces within the knee, in order to alleviate the major source of pain.

Although total knee arthroplasty is an established surgical treatment option, up to 20% of patients may be dissatisfied with the outcome , and many prostheses fail over time, requiring costly revision surgery. Current understanding suggests that soft tissue balancing has a crucial role to play in the outcome of total knee arthroplasty. Instability after total knee replacement is an important cause of failure. It is not clear what the normal collateral ligament laxity should be. There is a paucity of current data on normal knee collateral ligament laxity . Nevertheless, restoring this may improve patient satisfaction with TKA and longevity. It appears that there is considerable variation between individuals, genders , and ethnic groups , when it comes to "normal" laxity. However, much of the existing data relates to healthy young volunteers , and it is not clear how this information should map against the elderly osteoarthritic population who are most likely to be in need of TKA. Recent advances in computer assisted navigation have provided surgeons with a more precise measure of knee alignment , and knee laxity .

Orthopaedic surgeons at New Cross Hospital have been utilising this technology to improve intraoperative placement of total knee replacement implants since 2015. Computer navigation is carried out using the Stryker Precision Navigation System. This system records kinematic and static measurements of knee alignment and laxity in patients just prior to the commencement of the total knee replacement procedure.

By gathering and analysing data from this machine, on the degree of laxity in osteoarthritic patients about to undergo TKA, I this study aims to gain a greater understanding of what can be considered "normal" and whether there are significant differences between individuals, and between ethnic populations in this regard. This will help future surgical decision making about how tight or loose prosthetic knee replacements should be, based on individual characteristics.

ELIGIBILITY:
Inclusion Criteria:

* All cases of TKA recorded on the 2 Stryker navigation machines based at New Cross and Cannock Chase Hospitals will be included in the study. Duplicates will be identified and removed from the case series.

Exclusion Criteria:

* Cases in which there is incomplete or inadequate kinematic data recorded in the machine database will be excluded from the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing total knee arthroplasty between 2015 and 2019 under the care of a single Consultant
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The degree of ligamentous laxity in severely arthritic knees | 4 weeks
  kinematic and static measurements pre and post op laxity in flexion and extension
Pattern of laxity in relation to pre-existing knee deformity | 4 weeks
  Establish a pattern of laxity in relation to pre-existing knee deformity
Baseline ligamentous laxity between males and females, and between Caucasian and Asian populations | 4 weeks
  To compare baseline ligamentous laxity between males and females, and between Caucasian and Asian populations

CONTACTS AND LOCATIONS:
Overall Officials: George Hirsch, Study Director — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No